CLINICAL TRIAL: NCT05905055
Title: A Phase 3, Multi-Center, Randomized, Single-Blind Study to Assess the Efficacy and Safety of Cefepime/Nacubactam and Aztreonam/Nacubactam Versus Best Available Therapy in Adults With Complicated Urinary Tract Infection, Acute Uncomplicated Pyelonephritis, Hospital-Acquired Bacterial Pneumonia, Ventilator Associated Bacterial Pneumonia, and Complicated Intra-Abdominal Infection Due to Carbapenem Resistant Enterobacterales
Brief Title: P3 Study to Assess Efficacy and Safety of Cefepime/Nacubactam and Aztreonam/Nacubactam Versus Best Available Therapy for Adults With Infection Due to Carbapenem Resistant Enterobacterales
Acronym: Integral-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP0595-6
Record Dates: First submitted 2023-03-02; First posted 2023-06-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis; Hospital-acquired Bacterial Pneumonia; Ventilator-associated Bacterial Pneumonia; Complicated Intra-abdominal Infection
Keywords: nacubactam; OP0595; Integral-2
MeSH Terms: interventions — nacubactam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- co-administration of cefepime and nacubactam (Experimental): co-administration of 2 g cefepime and 1 g nacubactam q8h (60 min. infusion)
  Interventions: Drug: co-administration of cefepime and nacubactam
- co-administration of aztreonam and nacubactam (Experimental): co-administration of 2 g aztreonam and 1g nacubactam q8h (60 min. infusion)
  Interventions: Drug: co-administration of aztreonam and nacubactam
- BAT (Active Comparator): Best Available Therapy
  Interventions: Drug: BAT

INTERVENTIONS:
Drug: co-administration of cefepime and nacubactam — 2 g cefepime and 1 g nacubactam every 8 hours for at least 5 days and up to 14 days via IV infusion over a period of 60 minutes
  Arms: co-administration of cefepime and nacubactam
Drug: co-administration of aztreonam and nacubactam — 2 g aztreonam and 1 g nacubactam every 8 hours for at least 5 days and up to 14 days via IV infusion over a period of 60 minutes
  Arms: co-administration of aztreonam and nacubactam
Drug: BAT — Dosage of BAT will be based per site's standard of care
  Arms: BAT

SUMMARY:
This study is a multi-center, randomized, single-blind, parallel-group study to assess the efficacy and safety, when nacubactam is coadministered with cefepime or aztreonam, compared with best available therapy (BAT), in the treatment of patients with cUTI, AP, HABP, VABP, and cIAI, due to Carbapenem Resistant Enterobacterales.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients at least 18 years of age (or age of legal consent, whichever is older) at the time of obtaining informed consent and who can be hospitalized throughout the Treatment Period;
2. Weight at most 140 kg;
3. The following criteria must be satisfied:

   a. For known CRE infection, meets either of the following (i or ii): i. Has a known CRE infection, alone or as a single isolate of a polymicrobial infection, based on evidence from CRE culture, susceptibility testing, and possible carbapenemase phenotypic testing (or possible molecular testing) within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug; AND Has received no more than 24 hours of an antimicrobial agent to which the known CRE is known to be susceptible within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug; OR ii. Has a known CRE infection, alone or as a single isolate of a polymicrobial infection, based on evidence from CRE culture, susceptibility testing, and possible carbapenemase phenotypic testing (or possible molecular testing) within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug; AND Has documented clinical evidence of failure (ie, clinical deterioration or failure to improve) after at least 48 hours of treatment with an antimicrobial agent to which the known CRE is known to be susceptible within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug; b. For suspected CRE infection, meets the following (i or ii): i. Has a suspected CRE infection, alone or as a single isolate of a polymicrobial infection, based on evidence which may be determined within 90 days prior to the first dose of study drug through rapid diagnostic tests, active surveillance cultures, other documentation of CRE colonization, or prior infection due to a CRE pathogen; AND Has received no more than 24 hours of empiric antimicrobial therapy for Gram negative organisms within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug； ii. Has a suspected CRE infection, alone or as a single isolate of a polymicrobial infection, based on evidence which may be determined within 90 days prior to the first dose of study drug through rapid diagnostic tests, active surveillance cultures, other documentation of CRE colonization, or prior infection due to a CRE pathogen; AND Has documented clinical evidence of failure (ie, clinical deterioration or failure to improve) after at least 48 hours of treatment with empiric antimicrobial therapy for Gram-negative organisms within 72 hours (or 96 hours for cIAI) prior to the first dose of study drug; Note: CRE is defined as Enterobacterales by susceptibility data of MIC at least 2 microg/mL to imipenem or meropenem OR imipenem or meropenem disk diffusion (zone diameter < 22 mm). If MIC or disk diffusion data are not available in the local laboratory or before the availability of MIC or disk diffusion results, each site can use other methods and criteria in the institution (eg, phenotypic or molecular testing) as the initial evidence of CRE for enrollment. In any case, pathogen identification and susceptibility testing performed at the central laboratory will be used to determine CRE in the final study analysis.

Exclusion Criteria:

1. Has a history of serious allergy, hypersensitivity (eg, anaphylaxis), or any serious allergic reaction to carbapenems, cephems, penicillins, other beta-lactam antibiotics, or any BLIs (eg, tazobactam, sulbactam, or clavulanic acid)
2. Has known or suspected single or concurrent infection with Acinetobacter spp., metallo-β-lactamase (MBL) producing Pseudomonas aeruginosa, or other organisms that are not adequately covered by the study drug (eg, concurrent viral, mycobacterial, or fungal infection) and need to be managed with other anti-infectives; Note: Patients with qualifying Gram-negative pathogen co-infected with a Gram-positive pathogen may be administered narrow spectrum, open-label glycopeptide (eg, vancomycin), oxazolidinone (eg, linezolid), or daptomycin concomitantly with the study drug at the discretion of the Investigator. Patients with cIAI may receive metronidazole in addition to cefepime/nacubactam, aztreonam/nacubactam, or as part of BAT if anaerobic coverage is deemed necessary
3. Has only a Gram-positive organism pathogen isolated from study-qualifying culture;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-09-22 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the proportion of patients with overall treatment success at TOC across all infection types (ie, cUTI, AP, HABP, VABP, and cIAI), which is a composite endpoint derived from the efficacy outcomes of each infection type. | 7 [±2] days after EOT [Day 10 to 23]
  For cUTI and AP, the composite clinical outcome of cure and the microbiological outcome of eradication are defined as the outcome of cure.
  For HABP and VABP, the clinical success is defined as the outcome of cure. For cIAI, the clincal success is defined as the outcome of cure.

CONTACTS AND LOCATIONS:
Locations (1):
- Meiji Research Site, Nankoku, Kochi, Japan